CLINICAL TRIAL: NCT05332613
Title: Diet and Meal Timing in Patients With Non-Alcoholic Fatty Liver Disease: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-10024103
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Trehalase

STUDY DESIGN:
Intervention Model Description: This is a single-site, randomized, controlled pilot study. The investigators hypothesize that time-restricted eating (TRE) will lead to an additional improvement in hepatic steatosis as compared to standard of care lifestyle recommendations alone measured by MRI-PDFF. The investigators plan to enroll 40 participants to two arms between the years of 18 and 65 with NAFLD as defined by MRI-PDFF score of greater or equal to 10%. Participants on the experimental arm (TRE plus SOC) will be required to fast for 16 hours each day for 12 weeks. Counseling will involve instructing the participant to choose an 8-hour eating window. During the fasting window, the participant is able to drink water and black coffee or tea. Participants in both arms will be given lifestyle recommendations with respect to diet and exercise. The RD will instruct participants regarding standard of care lifestyle recommendations, which includes education of a low-calorie diet and moderate-intensity exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TRE plus SOC (Experimental): Participants will be required to fast each day for 12 weeks and will be given lifestyle recommendations with respect to diet and exercise. The registered dietitian (RD) will obtain a baseline dietary record and provide counseling on the time-restricted eating regimen. The RD will collect the participant's normal diet and exercise routine. Counseling will involve instructing the participant to choose an eight-hour eating window (e.g., 10:00am - 6:00pm) during which the participant will be able to eat. During the 16-house fasting window (e.g., 6:00pm - 10:00 am), the participant is able to drink regular water and black coffee or tea. The RD will be available to answer any questions the participants may have pertaining to the regimen and will instruct the participants regarding standard of care lifestyle recommendations. This includes education of a low-calorie diet (500-1000 kcal) and moderate-intensity exercise.
  Interventions: Behavioral: TRE plus SOC
- SOC (Active Comparator): lifestyle modifications and weight management. Participants will be given lifestyle recommendations with respect to diet and exercise. The registered dietitian (RD) will obtain a baseline dietary record and provide counseling on the time-restricted eating regimen. A baseline dietary record will be assessed prior to fasting initiation with the RD in person. The RD will also collect the subject's normal diet and exercise routine. The RD will instruct the participants regarding standard of care lifestyle recommendations. This includes education of a low-calorie diet (500-1000 kcal) and moderate-intensity exercise.
  Interventions: Behavioral: SOC
- Crossover to TRE (Experimental): Participants who have not lost weight or have lost less than or equal to 5% of their body weight, they will be given the option to crossover to the TRE arm. Following the initial 12-week period and end of study MRI, participants would restart another identical 12-week cycle but adhering to the exact steps of the TRE arm including another 4 visits with the registered dieticians (RDs) and an end of study visit with repeat Fibroscan, InBody 770 body composition scan, and MRI-PDFF.
  Interventions: Behavioral: TRE

INTERVENTIONS:
Behavioral: TRE plus SOC — Participants will undergo time restricted eating (TRE) each day for 12 weeks and will be given lifestyle recommendations with respect to diet (500-1000 kcal) and moderate-intensity exercise (30 minutes).
  Arms: TRE plus SOC
Behavioral: SOC — Participants will be given lifestyle recommendations with respect to diet (500-1000 kcal) and moderate-intensity exercise (30 minutes).
  Arms: SOC
Behavioral: TRE — Participants will undergo time restricted eating (TRE) each day for 12 weeks plus 4 extra visits with the registered dietician and repeat Fibroscan, InBody composition scan, and MRI-PDFF.
  Arms: Crossover to TRE

SUMMARY:
This study will assess the impact of time-restricted eating (8 hours of eating each day) with standard of care lifestyle recommendations (hypocaloric, Mediterranean diet and 30 minutes of exercise on at least 5 days/week) on the degree of fat in the liver as measured by magnetic resonance imaging.

DETAILED DESCRIPTION:
Time-Restricted Eating (TRE) is a form of caloric restriction through daily prolonged fasting that has been shown to lead to weight loss, improved glucose regulation, and suppression of inflammation. Non-alcoholic fatty liver disease (NAFLD) is a metabolic condition that in certain patients can lead to significant morbidity and mortality. The only current treatment for NAFLD is weight loss. In the proposed study, the investigators aim to test the hypothesis that TRE will add additional benefit in the treatment of NAFLD on top of standard of care diet and lifestyle modifications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 65 years old
* Must provide signed written informed consent and agree to comply with the study protocol
* BMI >25 kg/m²
* Baseline liver fat content of at least 10% as measured by MRI-PDFF

Exclusion Criteria:

* Unclear etiology of liver disease
* Competing etiologies for hepatic steatosis
* Co-existing causes of chronic liver disease according to standard diagnostic testing including, but not restricted to:
* Positive hepatitis B surface antigen
* Positive hepatitis C virus RNA
* Suspicion of drug-induced liver disease
* Alcoholic liver disease
* Autoimmune hepatitis
* Wilson's disease
* Hemochromatosis
* Primary biliary cholangitis or primary sclerosing cholangitis
* Known or suspected hepatocellular carcinoma
* Current or recent history (<5 years) of significant alcohol consumption. For men, significant consumption is defined as >30g of alcohol per day. For women, it is defined as >20g of alcohol per day.
* Compensated and decompensated cirrhosis (clinical and/or histologic evidence of cirrhosis). NASH patients with fibrosis stage = 4 according to the NASH CRN fibrosis staging system are excluded.
* Reduction in weight by ≥ 5% within the prior 90 days
* Current fasting for ≥ 12 hours per day on the majority of days each week
* Pregnant females
* Mental instability or incompetence, such that the validity of the informed consent or ability to be compliant with the study is uncertain
* Inability to perform MRI-PDFF and/or study as defined below
* Inability to medically perform prolonged fasting (i.e. insulin regimen)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients Who Achieve At Least 30% Reduction in Liver Fat at 12 Weeks | 12 weeks
  Evaluate the percentage of patients with baseline NAFLD (MRI-PDFF greater than or equal to 10%) who achieve clinically significant improvement in hepatic fat, as defined by greater than or equal to 30% reduction from baseline liver fat on MRI-PDFF, while adopting a time-restricted eating pattern (fasting 16 hours per day) along with standard of care management as compared to patients with only standard of care NAFLD management.

SECONDARY OUTCOMES:
Mean Change from Baseline in Quality of Life Score on SF-36 at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change of quality of life score from SF-36 from baseline to 12 weeks. Scores range from 0-100. Higher scores indicate better health status, while lower scores indicate a poorer health status. A mean score of 50 has been articulated as the normative value of all scales.
Mean Change from Baseline in Weight at 12 weeks | Baseline, 12 weeks
Mean Change from Baseline in BMI at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change of body mass index from baseline to 12 weeks.
Mean Change from Baseline in Liver Stiffness on Fibroscan® at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change in liver stiffness as measured by (FibroScan®) from baseline to 12 weeks.
Mean Change from Baseline in Body Composition Measurements at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change of body composition measurements as measure by InBody Body
Mean Change from Baseline in aspartate transglutaminase at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change in aspartate transglutaminase from baseline to 12 weeks.
Mean Change from Baseline in alanine transglutaminase at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change in alanine transglutaminase from baseline to 12 weeks.
Mean Change from Baseline in total bilirubin at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change in total bilirubin from baseline to 12 weeks.
Mean Change from Baseline in direct bilirubin at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change direct bilirubin from baseline to 12 weeks.
Mean Change from Baseline in albumin at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change in albumin from baseline to 12 weeks.
Mean Change from Baseline in total protein at 12 weeks | Baseline, 12 weeks
  Evaluate the mean change in total protein from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sonal Kumar, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No